CLINICAL TRIAL: NCT00606983
Title: Prevention of Acute Voiding Difficulty After Radical Proctectomy for Rectal Cancer With Tamsulosin
Brief Title: Prevention of Acute Voiding Difficulty After Radical Proctectomy
Status: Completed | Phase: Phase 3 | Type: Interventional
Sponsor: Seoul National University Hospital (Other)
Responsible Party: Sung-Bum Kang, Department of Surgery, Seoul National University Bundang Hospital
Allocation: Randomized | Model: Parallel | Masking: Triple | Purpose: Treatment
Other Study IDs: B-0702-042-006; SNUBH-GS-CR3
Record Dates: First submitted 2008-01-22; First posted 2008-02-05 (Estimated); Last update posted 2011-07-20 (Estimated); Status verified 2011-07

CONDITIONS: Rectal Cancer; Urinary Retention
MeSH Terms: conditions — Rectal Neoplasms; Urinary Retention | interventions — Tamsulosin

STUDY DESIGN:
Who Masked: Participant, Care Provider, Investigator
Oversight: Data Monitoring Committee: Yes

ARMS (2):
- 1 (No Intervention)
- 2 (Experimental): oral administration of Tamsulosin
  Interventions: Drug: Tamsulosin

INTERVENTIONS:
Drug: Tamsulosin — oral administration of Tamsulosin
  Arms: 2

SUMMARY:
Various adrenergic blockers are used for acute voiding difficulty after proctectomy. Recently, a selective alpha5-adrenergic blocker, Tamsulosin has been reported to have benefit in reducing urinary symptom score and in reducing the rate of intermittent self-catheterization for patients with rectal cancer after radical proctectomy.

This study is to evaluate the efficacy of pharmacologic prevention to ameliorate the incidence of postoperative urinary dysfunction.

DETAILED DESCRIPTION:
Acute voiding difficulty is caused from damage to pelvic sympathetic nerve after rectal surgery, and usually resolved spontaneously within several months after the surgery. However, acute voiding difficulty results in prolonged insertion of urinary catheter and is associated risk for urinary tract infection. Various adrenergic blockers are used for acute voiding difficulty after proctectomy. Recently, a selective alpha5-adrenergic blocker, Tamsulosin has been reported to have benefit in reducing urinary symptom score and in reducing the rate of intermittent self-catheterization for patients with rectal cancer after radical proctectomy.

This study is to evaluate the efficacy of pharmacologic prevention to ameliorate teh incidence of postoperative urinary dysfunction.

ELIGIBILITY:
Inclusion Criteria:

* Patients between 20-80 years old in general good health
* Patient willing to participate in the study
* Patient who understands and accepts to sign the informed consent form
* Patient who received proctectomy for rectal cancer located 15 cm or less of the anal verge

Exclusion Criteria:

* Documented problem of preoperative urinary dysfunction
* Any post-surgery change in patient condition which requires insertion of urinary catheter after surgery
* Past history of recurrent urinary tract infection or malignancy of urinary system organs
* Past history of surgery for urinary system organs
* Current administration of Finasteride or Dutasteride
* Liver dysfunction (SGOT or SGPT 100 IU/L or more)
* Kidney dysfunction (serum Creatinine 3mg/dl or more)

Ages: 20 Years to 80 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 100 (Estimated)
Dates: Start 2007-05; Primary Completion 2010-09 (Actual); Study Completion 2010-09 (Actual)

PRIMARY OUTCOMES:
Re-insertion rate of urinary catheter after removal | after removal of urinary catheter

SECONDARY OUTCOMES:
Scores of IPSS (International Prostatic Symptom Score) and the results of uroflowmetry | at postoperative day 7

CONTACTS AND LOCATIONS:
Overall Officials: Sung-Bum Kang, M.D., Ph.D, Principal Investigator — Seoul National University Bundang Hospital
Locations (1):
- Department of Surgery, Seoul National University Bundang Hospital, Seongnam, South Korea

REFERENCES:
- [Derived] Ellahi A, Stewart F, Kidd EA, Griffiths R, Fernandez R, Omar MI. Strategies for the removal of short-term indwelling urethral catheters in adults. Cochrane Database Syst Rev. 2021 Jun 29;6(6):CD004011. doi: 10.1002/14651858.CD004011.pub4. PMID 34184246